CLINICAL TRIAL: NCT03082781
Title: A Comparative Assessment of Weight Loss and Anti-lipid Effects of Negative Calorie Diet and Low-calorie Diet in Overweight/Obese Middle-aged and Older Women Under Exercise Condition
Brief Title: Dietary Choice in Active Older Adult Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: P.L.Shupik National Medical Academy of Post-Graduate Education (Other)
Responsible Party: Principal Investigator, Mohammadreza Rezaeipour, MD, PhD, Asst. Prof. of sports medicine (sports injury and corrective movement), University of Sistan and Baluchestan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: No Grant 5
Record Dates: First submitted 2017-03-05; First posted 2017-03-17 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Exercise Addiction; Diet Habit; Obesity; Overweight; Weight Loss
Keywords: Diet; Exercise; Obesity; Overweight; Weight loss
MeSH Terms: conditions — Feeding Behavior; Obesity; Overweight; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group I (Experimental): Study group I (57 participants) received the NCD with exercise (NCDsport).This groups had 5% caloric restriction from their maintenance energy requirements and 10% increase in energy expenditure through structured regular exercise.
  Interventions: Dietary Supplement: NCDsport
- Study group II (Experimental): Study group II (54 participants) received the low-calorie diet with exercise (LCDsport). This groups had 5% caloric restriction from their maintenance energy requirements and 10% increase in energy expenditure through structured regular exercise.
  Interventions: Dietary Supplement: LCDsport

INTERVENTIONS:
Dietary Supplement: NCDsport — Negative Calorie Diet supplemented with exercise
  Other Names: group I
  Arms: Study group I
Dietary Supplement: LCDsport — Low-Calorie diet with exercise
  Other Names: group II
  Arms: Study group II

SUMMARY:
The present study aimed to determine the effects of negative-calorie diet supplemented with exercise, on weight loss and lipid profile, and to compare its efficiency with low-calorie diet with exercise among elderly adult women with abnormal weight gain.

DETAILED DESCRIPTION:
Background: Negative-calorie diet is among the popular dieting guides for weight loss; however, there is still little knowledge about this method.

Objectives: The present study aimed to determine the effects of negative-calorie diet supplemented with exercise, on weight loss and lipid profile, and to compare its efficiency with low-calorie diet with exercise among elderly adult women with abnormal weight gain.

Material and Methods: Participants included sedentary women (age 45-75 years) with overweight or obesity (n=111). They were randomly divided into two groups including negative calorie diet with exercise, and low-calorie diet with exercise. Of all 111 participants, 90 persons completed the treatment. The weight assessment parameters including change in weight and body composition, blood sample tests were performed pre- and three month post-intervention.

ELIGIBILITY:
Inclusion Criteria:

Non-smokers and weight-stable (± 2 kg, for more than one year) with no history of regular exercise in at least three months before the study.

Exclusion Criteria:

History of CVD and other disorders such as diabetes, depression, eating disorders, chronic medications, kidney disease, cancer, food allergies or intolerances to items used in meals. Subjects with abnormality in thyroid or Electrocardiograph, any history of anti-obesity medication or weight loss drugs or dietary supplementations for weight control.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants were non-smokers and weight-stable (± 2 kg, for more than one year) with no history of regular exercise in at least three months before the study.
Enrollment: 66 (Actual)
Dates: Start 2012-10-10 (Actual); Primary Completion 2013-06-20 (Actual); Study Completion 2013-08-15 (Actual)

PRIMARY OUTCOMES:
Weight | Baseline
  assessed in kg
Total cholesterol (Total-C) | Baseline
  assessed in mg/dl
High-density lipoprotein -cholesterol (HDL-C) | Baseline
  assessed in mg/dl
Low-density lipoprotein -cholesterol (LDL-C) | Baseline
  assessed in mg/dl
Triglycerides (TG) | Baseline
  assessed in mg/dl

SECONDARY OUTCOMES:
Weight | 3-month
  assessed in kg
Total cholesterol (Total-C) | 3-month
  assessed in mg/dl
High-density lipoprotein -cholesterol (HDL-C) | 3-month
  assessed in mg/dl
Low-density lipoprotein -cholesterol (LDL-C) | 3-month
  assessed in mg/dl